CLINICAL TRIAL: NCT04649502
Title: Rediscovery of Metformin for the Chronic Disabling Auto-inflammatory Disease Hidradenitis Suppurativa
Brief Title: Metformin for the Treatment of Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: K.R. van Straalen (Other)
Responsible Party: Sponsor-Investigator, K.R. van Straalen, MD., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMCD20022
Record Dates: First submitted 2020-11-16; First posted 2020-12-02 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin combined with doxycycline (Experimental)
  Interventions: Combination Product: Metformin
- Doxycyline combined with placebo (Placebo Comparator)
  Interventions: Combination Product: Metformin

INTERVENTIONS:
Combination Product: Metformin — Metformin in combination with doxycycline

SUMMARY:
A randomized controlled trial investigating the metformin is the treatment for hidradenitis suppurativa. Metformin combined with doxycycline will be compared to the standard treatment of doxycycline monotherapy for HS severity and the effect on the pre-diabetic condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at baseline
* A diagnosis of HS for at least 1 year prior to baseline
* mild to moderately active disease defined by a HS Physician Global Assessment (HS-PGA) score of 2-3 and the Refined Hurley classification of mild to moderate at baseline
* Indication for systemic therapy; i.e. uncontrolled disease under conventional topical therapy.
* Able and willing to give written informed consent and to comply with the study requirements

Exclusion Criteria:

* Pregnant and lactating women
* Concomitant diabetes mellitus
* Use of antibiotics within 14 days prior to baseline
* Use of immunosuppressing/modulating therapies within 28 days prior to baseline
* A known allergy to metformin or doxycycline or any of the ingredients metformin or doxycycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
IHS4 | 24 weeks
  International Hidradenitis Suppurativa Severity Score System (IHS4)

SECONDARY OUTCOMES:
Insulin resistance | 12 and 24 weeks
  • Change in insulin resistance from baseline using the HOMA-IR (based on fasting glucose and insulin levels) and differences between the groups at week 12 and 24.
Lesion Count | 12 and 24 weeks
  • Change in lesion count from baseline and differences between the groups at 12 and 24 week. Difference in lesion count will be assessed between the groups at week 12 and 24.
NRS-Pain | 12 and 24 weeks
  Change in skin related pain from baseline, on a numerical rating scale, and differences between the groups at week 12 (V2) and 24 (V4)
Cost-effectiveness | 24 weeks
  • For cost-effectiveness the direct medical costs will be will be assessed using the iMTA Medical Consumption Questionnaire (iMCQ), The measurement will be at baseline, at 12 weeks and at 24 weeks. Productivity losses will be collected using the iMTA Productivity Cost Questionnaire (iPCQ) includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work. The friction cost method for valuing the production losses will be applied in accordance to the Dutch manual for costing studies. Hence, the productivity loss will be valued per worker by age and gender and, for long term absences, taking into account that productivity costs to society is confined to the period needed to replace a worker (the friction period). Cost effectiveness will be estimated using Dutch manual for costing studies in economic evaluations (publication of the Health Care Institute (ZIN).
Bio-markers | 24 weeks
  * The correlation between baseline calprotectin levels and disease severity for both groups.
  * The correlation between calprotectin levels and treatment response in each group at week 12 and 24.
Safety and Tolerability | up to 24 weeks
  • Incidence and severity of all adverse events (according to medDRA) will be analysed throughout the study, and renal function and lactate will be assessed at every visit.
Metabolic syndrome | 12 and 24 weeks
  Change in parameters of metabolic syndrome (waist circumference, blood pressure, HDL cholesterol, and triglycerides) from baseline and differences between the groups at week 12 and 24.
Pre-diabetic disorder | 12 and 24 weeks
  Change in HbA1c from baseline and differences between the groups at week 12 and week 24.
HiSCR | 12 and 24 weeks
  The percentage of HiSCR achievers (a ≥ 50% reduction in inflammatory lesion count (abscesses + inflammatory nodules), and no increase in abscesses or draining fistulas when compared with baseline) and the difference between the groups at week 12 and 24.
HS-PGA | 12 and 24 weeks
  The change in HS-PGA from baseline and the difference between the groups at week 12 and 24.
Flares | 12 and 24 weeks
  Change in self-reported frequency of flares from baseline and differences between the groups at week 12 and 24.
DLQI | 12 and 24 weeks
  Change in quality of life from baseline and differences between the groups, measured with the Dermatologic Life Quality Index and the EQ-5D, at week 12 and 24.
Treatment satisfaction | up to 24 weeks
  Difference in treatment satisfaction and recommendation on a 5- and 3-point Likert scale respectively at week 12 and 24 between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided